CLINICAL TRIAL: NCT00622024
Title: Perioperative Depression and Postoperative Arrhythmia in Elective Coronary Bypass Graft Surgery
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB#06-0116-AE
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Artery Disease
Keywords: Arrhythmia; Depression; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Arrhythmias, Cardiac; Depression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative arrhythmias (heart irregularities) are one of the most common complications after cardiac surgery and are associated with increased morbidity and mortality. Preoperative depression may be an important co-factor in the generation of postoperative arrhythmias due to sympathetic hyperactivity evident in patients with depression.

Objectives: To determine the effect of preoperative depression on postoperative arrhythmia in patients undergoing elective coronary artery bypass graft (CABG) surgery.

Prospective observational study, 120 patients undergoing elective CABG surgery ECG will be preformed preoperatively on all patients. All patients will be assessed for signs of depression using the Prime MD Patient Health Questionnaire (Prime MD PHQ) one week before surgery and 6 weeks postoperatively.Based on the Prime MD PHQ results, patients will be divided into two groups: those with or without signs of depression. Heart rate and rhythm monitoring with Holter will be performed for 3 days postoperatively in order to compare the incidence of postoperative arrhythmias between groups.

The primary outcome is the number of patients with and without depression suffering from ventricular and/or supraventricular arrhythmias. Secondary outcomes include all cause mortality, non-fatal myocardial infarction, cardiac arrest, and congestive heart failure.

CABG surgery is the most common operative procedure in North America and arrhythmias are one of the most common postoperative complication. It is estimated that about a third of these cardiac patients suffer from preoperative depression and therefore may be exposed to a higher risk of perioperative morbidity and mortality. If an association between preoperative depression and postoperative arrhythmia is found, treatment modalities may be indicated to reduce the prevalence of perioperative arrhythmia in patients with preoperative depression undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-75 years of age undergoing elective CABG surgery.
* Patients must provide informed consent

Exclusion Criteria:

* Patients with a history of arrhythmias (AF, supraventricular tachycardia, ventricular tachycardia, ventricular fibrillation, permanent pacemaker and/or defibrillator).
* Patients who are unable to read.
* Patients with significant psychiatric disorders other than depression.
* Patients with a history of pulmonary hypertension.
* Patients with a left ventricular ejection fraction < 40%.
* Patients with cognitive impairment as measured by the MMSE.
* Patients on antidepressants at the time of assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective CABG surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with and without depression suffering from ventricular and/or supraventricular arrhythmias | Depression assessment and holter monitor 3days postop

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — Toronto General Hospital, UHN
Locations (1):
- Toronto General Hospital, UHN, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Katznelson R, Scott Beattie W, Djaiani GN, Machina M, Lavi R, Rao V, Lavi S. Untreated preoperative depression is not associated with postoperative arrhythmias in CABG patients. Can J Anaesth. 2014 Jan;61(1):12-8. doi: 10.1007/s12630-013-0051-3. Epub 2013 Nov 12. PMID 24218191